CLINICAL TRIAL: NCT01117792
Title: Subcutaneous Implantable Defibrillator (S-ICD) System - CE Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DN-01040
Record Dates: First submitted 2010-04-28; First posted 2010-05-05 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: ACC/AHA/NASPE Class 1, IIa or IIb Indications
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-ICD System (Experimental)
  Interventions: Device: subcutaneous implantable defibrillator (S-ICD) system

INTERVENTIONS:
Device: subcutaneous implantable defibrillator (S-ICD) system — implantable defibrillator system

SUMMARY:
The primary objective is to evaluate the S-ICD system's ability to identify and terminate induced ventricular fibrillation in patients during the implant procedure. The safety and performance of the S-ICD system will also be assessed throughout the patient follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Replacement of an existing implanted transvenous ICD system
* Class I, Class IIa, or Class IIb ACC/AHA/HRS indications for patients without an existing transvenous ICD system
* Age is >= 18 years
* Appropriate pre-operative ECG as measured with a specially developed template

Exclusion Criteria:

* Subjects unable or unwilling to provide informed consent
* Any condition which precludes the subject's ability to comply with the study requirements
* Females who are pregnant or lactating and pre-menopausal women who are unwilling to use adequate birth control for the duration of the study
* Participation in another investigational device trial at any time during the conduct of the S-ICD system trial without written consent from the sponsor.
* Patients with a serious medical condition and life expectancy of less than one year.
* Patients with documented spontaneous and frequently recurring VT that is reliably terminated with anti-tachycardia pacing
* Patients with existing epicardial patches or subcutaneous electrodes in the left thoracic quadrant
* Patients with impaired kidney function as measured by a Cockcroft-Gault Glomerular Filtration Rate (GFR) with a GFR <= 29.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen O'Connor, PhD, Hon FRCP, Study Director — Boston Scientific Corporation
Locations (8):
- Policlinico San Donato, San Donato Milanese, Italy
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum, Groningen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Russells Hall Hospital, Dudley, United Kingdom

REFERENCES:
- [Derived] Theuns DA, Crozier IG, Barr CS, Hood MA, Cappato R, Knops RE, Maass AH, Boersma LV, Jordaens L. Longevity of the Subcutaneous Implantable Defibrillator: Long-Term Follow-Up of the European Regulatory Trial Cohort. Circ Arrhythm Electrophysiol. 2015 Oct;8(5):1159-63. doi: 10.1161/CIRCEP.115.002953. Epub 2015 Jul 6. PMID 26148819

RESULTS

PARTICIPANT FLOW:
Groups:
- S-ICD System: Subjects enrolled and implanted with a Cameron Health subcutaneous implantable cardioverter defibrillator (S-ICD) system.
Period: Overall Study
Arm/Group | S-ICD System
Started | 55
Completed | 51
Not Completed | 4
Not completed — Death | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Subjects enrolled and implanted with a Cameron Health subcutaneous implantable cardioverter defibrillator (S-ICD) system.
Arm/Group | S-ICD System
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 34
  European | 9
  New Zealander, European | 8
  Maori | 2
  Indian | 1
  Asian | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 21
  Netherlands | 21
  Italy | 5
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Conversion of Induced Ventricular Fibrillation
Description: The total number of subjects the S-ICD System was successful at converting induced sustained ventricular fibrillation.
Time Frame: Testing done during the implant procedure
Population: Investigator induce sustained ventricular fibrillation conversion efficacy. Two of the 55 subjects implanted did not induce sustained ventricular fibrillation leaving 53 evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | S-ICD System
Number analyzed (Participants) | 53
Participants | 52

ADVERSE EVENTS:
Arm/Group | S-ICD System
All-Cause Mortality (participants affected / at risk) | 1/55
Serious Adverse Events (participants affected / at risk) | 17/55
Other Adverse Events (participants affected / at risk) | 4/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-ICD System (N=55)
Other - Adverse Event Terms Unknown (General disorders) | 17 (22)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-ICD System (N=55)
Other - Adverse Event Terms Unknown (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There is NOT an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.